CLINICAL TRIAL: NCT00990860
Title: START (Study in Asia of the Combination of Transcatheter Arterial Chemoembolization (TACE) With Sorafenib in Hepatocellular Carcinoma (HCC) Patients) Trial
Brief Title: Study in Asia of the Combination of TACE With Sorafenib in HCC Patients
Acronym: START
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Yee Chao, Taipei Veterans General Hospital,Taiwan
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ISS-13967; ISS-13967
Record Dates: First submitted 2009-09-01; First posted 2009-10-07 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Combination of TACE With Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Experimental)
  Interventions: Drug: doxorubicin; Procedure: TACE (Transcatheter arterial chemoembolization)

INTERVENTIONS:
Drug: doxorubicin — After identifying the target artery of HCC, doxorubicin will be infused through the target artery of HCC patient with lipiodol emulsion (dependent on the tumor size)
Procedure: TACE (Transcatheter arterial chemoembolization) — TACE (Transcatheter arterial chemoembolization)

SUMMARY:
TACE possibly plays a significant role in contributing to a subgroup of surviving residual tumor tissue which is characterized by more aggressive biology. This explains the strong scientific rationale for exploring the role of anti-angiogenic therapy such as sorafenib to remedy and strengthen the therapeutic efficacy of TACE to combat liver cancers. Sorafenib plays a prominent auxiliary role by further suppressing the tumor growth and prolonging the time to recurrence and progression. Performing TACE under sorafenib administration may have synergic effect on hepatic tumoral lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18
* life expectancy > 12 weeks
* Histologically diagnosed HCC, OR clinically diagnosed HCC for patients with difficulty in obtaining histological diagnosis. A clinically diagnosed HCC should fulfill ALL the criteria below

  * Chronic hepatitis B or C and/or evidence of liver cirrhosis.
  * Presence of hepatic tumour(s) with image findings compatible with HCC, and no evidence of other gastrointestinal tumours
  * A persistent elevation of serum AFP >= 400 ng/ml without any evidence of an existing α-fetoprotein-secreting germ cell tumour
* Child-Pugh score ≦ 7
* BCLC B
* The patient must have a solitary hepatic tumour greater than 3 cm in diameter or multifocal disease as evidenced by CT or MRI scanning.
* The target lesion must not have been previously treated with local therapy
* The patient must not be a candidate for surgical resection or ablation of the tumour. Size of largest tumor ≦10cm in largest dimension
* Patients who have received previous local therapy treatments (RFA, PEI, cryoablation, surgery, resection) to non-target lesions are eligible
* Local therapy must have been completed at least 4 weeks prior to baseline scan.
* ECOG performance status 0 or 1
* Hb ≧ 9g/dL,
* Absolute neutrophil count > 1000/mm3
* Platelet count ≧ 60x109/L
* Adequate clotting function: INR < 1.5
* Hepatic: AST or ALT < 5 X ULN
* Renal: serum creatinine < 1.5 x ULN
* Bilirubin ≦ 3mg/dL
* The patient must give written, informed consent

Exclusion Criteria:

* Tumor factors

  * Presence of extrahepatic metastasis
  * Predominantly infiltrative lesion
  * Diffuse tumor morphology with extensive lesions involving both lobes.
* Vascular complications

  * Hepatic artery thrombosis, or
  * Partial or complete thrombosis of the main portal vein, or
  * Tumor invasion of portal branch of contralateral lobe, or
  * Hepatic vein tumor thrombus, or
  * Significant arterioportal shunt not amenable to shunt blockage
* Liver function

  * Advanced liver disease: ascites, hepatic encephalopathy
  * Patients with clinically significant gastrointestinal bleeding within the 30 days prior to study entry.
* Others

  * Pregnant or lactating women.
  * Active sepsis or bleeding.
  * Hypersensitivity to intravenous contrast agents.
  * The patient has received prior treatment for HCC target lesion.
  * History of cardiac disease

    * Congestive heart failure > NYHA class 2; active coronary artery disease
    * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management.
  * Therapeutic anticoagulation with coumarin, heparins, or heparinoids.
  * Serious non-healing wounds (including wounds healing by secondary intention), acute or non-healing ulcers, or bone fractures within 3 months.
  * Impairment of swallowing that would preclude administration of sorafenib.
  * The patient is, in the opinion of the investigator, unable and / or unwilling to comply with treatment and study instructions.
  * Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted
  * Any active clinically serious infections (> grade 2 NCI-CTCAE ver 3.0)
  * HIV infection or AIDS-related illness or serious acute or chronic illness (based on medical history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability (such as adverse events and laboratory changes (haematology, clinical chemistry)) | 2 years

SECONDARY OUTCOMES:
Time to Progression | 2 years
Overall survival | 2 years
Progression Free Survival | 2 years
No. of TACE cycles | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yee Chao, Principal Investigator — VGH-TPE
Locations (8):
- Taiwan (8):
  - E-Da hospital, Kaohsiung City
  - Veterans General Hospital- Kaochiung, Kaoshiung
  - Veterans General Hospital- Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - Tri- Service General Hospital, Taipei
  - Veterans General Hospital- Taipei, Taipei
  - Chang-Gung Memorial Hospital- LinKou, TaoYuan Hsien

REFERENCES:
- [Derived] Chao Y, Chung YH, Han G, Yoon JH, Yang J, Wang J, Shao GL, Kim BI, Lee TY. The combination of transcatheter arterial chemoembolization and sorafenib is well tolerated and effective in Asian patients with hepatocellular carcinoma: final results of the START trial. Int J Cancer. 2015 Mar 15;136(6):1458-67. doi: 10.1002/ijc.29126. Epub 2014 Sep 16. PMID 25099027